CLINICAL TRIAL: NCT05184699
Title: The Effect of Dietary Intervention on Endothelial Glycocalyx Integrity and Microvascular Perfusion in Patients With Psoriatic Disease
Brief Title: The Effect of Dietary Intervention on Endothelial Glycocalyx in Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Professor of Cardiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 672/2-12-2021
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Psoriasis
Keywords: psoriasis; endothelial glycocalyx; arterial stiffness; coronary microcirculation; left ventricular myocardial deformation
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Sixty patients with psoriatic disease will be randomized to receive food supplement Endocalyx (n=30) or placebo (n=30) for 4 consecutive months.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food supplement Endocalyx (Active Comparator): Thirty patients with psoriatic disease will randomized to receive 4 capsules a day of the food supplement Endocalyx for 4 months
  Interventions: Dietary Supplement: Food supplement Endocalyx
- Placebo (Placebo Comparator): Thirty patients with psoriatic disease will randomized to receive 4 capsules a day of the placebo for 4 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Food supplement Endocalyx — Patients with psoriatic disease will be randomized to receive food supplement Endocalyx for 4 months.
  Other Names: Endocalyx; Q-prime
  Arms: Food supplement Endocalyx
Dietary Supplement: Placebo — Patients with psoriatic disease will be randomized to receive placebo for 4 months.
  Arms: Placebo

SUMMARY:
The food supplement Endocalyx is considered to support the endothelial glycocalyx integrity by supplying sulfated polysaccharides, anti-oxidant enzymes and additional substrates for glycocalyx synthesis. The investigators will study the effect of Endocalyx on endothelial, vascular and left ventricular myocardial function in patients with psoriatic disease.

DETAILED DESCRIPTION:
Sixty patients with psoriatic disease, who are referred to the outpatient psoriasis clinic of the Attikon University Hospital, will be randomized to receive food supplement Endocalyx (4 capsules per day) (n=30) or placebo (n=30) for 4 consecutive months.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian patients with psoriatic disease (plaque-type psoriasis or psoriatic arthritis)
* Body mass index ≥18.5 Kg/m2
* If female, patients must be non-pregnant and non-breastfeeding

Exclusion Criteria:

* History of acute coronary syndrome. Coronary artery disease will be excluded by a clinical history, examination and electrocardiogram.
* Moderate or severe valve disease
* Primary cardiomyopathies
* Chronic obstructive pulmonary disease
* Asthma
* Chronic kidney disease
* Liver failure
* Malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Endocalyx effects on endothelial glycocalyx thickness | four months
  Endocalyx effects on endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels using Sidestream Dark Field (SDF) imaging.

SECONDARY OUTCOMES:
Endocalyx effects on arterial stiffness | four months
  Endocalyx effects on arterial stiffness as assessed by carotid to femoral pulse wave velocity (PWV, m/s) using tonometry.
Endocalyx effects on coronary microcirculation | four months
  Endocalyx effects on coronary function as assessed by measuring coronary flow reserve of left anterior descending artery. Coronary flow reserve is estimated by Doppler echocardiography as the ratio of coronary flow velocity after bolus intravenous adenosine infusion to coronary flow velocity at rest.
Endocalyx effects on left ventricular myocardial function | four months
  Endocalyx effects on left ventricular function as assessed by global longitudinal strain using speckle-tracking echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Professor, Principal Investigator — 2nd Cardiology Department, National and Kapodistrian University of Athens
Locations (1):
- Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ikonomidis I, Katsanaki E, Thymis J, Pavlidis G, Lampadaki K, Katogiannis K, Vaiopoulos A, Lazarou V, Kostelli G, Michalopoulou E, Pililis S, Vlachomitros D, Theodoropoulos K, Vink H, Long R, Papadavid E, Lambadiari V. The Effect of 4-Month Treatment with Glycocalyx Dietary Supplement on Endothelial Glycocalyx Integrity and Vascular Function in Patients with Psoriasis. Nutrients. 2024 Aug 5;16(15):2572. doi: 10.3390/nu16152572. PMID 39125451